CLINICAL TRIAL: NCT06153251
Title: A Phase 1, Open-Label, Dose-Finding Study of BMS-986453, Dual Targeting BCMAxGPRC5D Chimeric Antigen Receptor T Cells, in Participants With Relapsed and/or Refractory Multiple Myeloma
Brief Title: A Study to Assess BMS-986453 in Participants With Relapsed and/or Refractory Multiple Myeloma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Juno Therapeutics, Inc., a Bristol-Myers Squibb Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA119-0002
Record Dates: First submitted 2023-11-22; First posted 2023-12-01 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Relapsed and/or Refractory Multiple Myeloma
Keywords: Dual Targeting; BCMAxGPRC5D; GPRC5DxBCMA; BMS-986453; CAR T; CART; Multiple Myeloma; Relapsed and/or Refractory
MeSH Terms: conditions — Multiple Myeloma | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Administration of BMS-986453 (Experimental)
  Interventions: Drug: BMS-986453; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: BMS-986453 — Specified dose on specified days
Drug: Fludarabine — Specified dose on specified days
Drug: Cyclophosphamide — Specified dose on specified days

SUMMARY:
The purpose of this study is to assess BMS-986453 in participants with relapsed and/or refractory multiple myeloma (RRMM).

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a diagnosis of multiple myeloma with relapsed and/or refractory disease.
* Participants must have confirmed progressive disease on or within 12 months (measured from the last dose) of completing treatment with the last anti-myeloma treatment regimen before study entry.
* Participants in Part A and Part B Cohort 1 and in Part B Cohort 2 must have relapsed/refractory multiple myeloma and received previous antimyeloma therapy, including a proteasome inhibitor and an immunomodulatory agent.
* Participants must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Participants must have adequate organ function.

Exclusion Criteria:

* Participants must not have any known active or history of central nervous system (CNS) involvement of multiple myeloma.
* Participants must not have active or history of plasma cell leukemia, Waldenstrom's macroglobulinemia, POEMS (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, skin changes) syndrome, or clinically significant amyloidosis.
* Participants must not have a history or presence of clinically significant CNS pathology such as seizure disorder, aphasia, stroke, severe brain injury, dementia, Parkinson's disease, or cerebellar disease, or presence of clinically active psychosis.

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-01-23 (Actual); Primary Completion 2030-05-02 (Estimated); Study Completion 2030-05-02 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-emergent adverse events (AEs) | Up to 4 years
Number of participants with serious adverse events (SAEs) | Up to 4 years
Number of participants with AEs leading to discontinuation | Up to 4 years
Number of participants with AEs leading to death | Up to 4 years
Number of participants with dose-limiting toxicities (DLTs) | Up to 4 years

SECONDARY OUTCOMES:
Maximum observed concentration (Cmax) | Up to 4 years
Time of maximum observed concentration (Tmax) | Up to 4 years
Area under the blood concentration-time curve from time zero to 28 days after dosing (AUC(0-28D)) | Up to 4 years
Overall response rate (ORR) | Up to 4 years
Complete response rate (CRR) | Up to 4 years
Number of participants with very good partial response (VGPR) or better | Up to 4 years
Progression-free survival (PFS) | Up to 4 years
Overall survival (OS) | Up to 4 years
Time to response (TTR) | Up to 4 years
Time to complete response (TTCR) | Up to 4 years
Duration of response (DOR) | Up to 4 years
Duration of complete response (DOCR) | Up to 4 years
Persistence of BMS-986453 in peripheral blood | Up to 4 years
  Defined as a transgene count greater than or equal to the lower limit of detection (LLOD)
Expansion rate | Up to 4 years
  Defined as Cmax divided by Tmax

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (19):
- United States (13):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - UCSF Helen Diller Medical Center at Parnassus Heights, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - Moffitt Cancer Center, Tampa, Florida
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Local Institution - 0008, Nashville, Tennessee
  - Tennessee Oncology, Nashville, Tennessee
  - Swedish Medical Center, Seattle, Washington
- Hôpital Saint-Louis, Paris, France
- Germany (3):
  - Universitaetsklinikum Koeln, Cologne
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Universitaetsklinikum Wuerzburg, Würzburg
- Spain (2):
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Hospital Universitario de Salamanca - Complejo Asistencial Universitario de Salamanca, Salamanca

IPD SHARING:
Plan to Share IPD: No
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myers Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-andresearch/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT06153251.html